CLINICAL TRIAL: NCT06172283
Title: A Pilot, Feasibility Study of Intermittent Fasting in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Brief Title: Intermittent Fasting in Prostate Cancer Patients Receiving Androgen Deprivation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Roberto Pili, Associate Dean for Cancer Research and Integrative Oncology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007635
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Longitudinal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intermittent Fasting (Experimental): Patients will undergo 16h periods of fasting everyday. Optionally, patients will be offered to undergo a plant-based diet consisting of 20% plant based protein, 50% carbohydrates, and 30% fat for the duration of the study.
  Interventions: Other: Intermittent Fasting

INTERVENTIONS:
Other: Intermittent Fasting — Dietary intervention

SUMMARY:
This is a a pilot study to assess the feasibility of intermittent caloric restriction (plus a plant-enriched diet optionally) in prostate cancer patients receiving androgen deprivation therapy. Study feasibility measures will include enrollment rate, drop-out rate and compliance with diet measured by self-reports.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation in this trial, the subject must:
* Be willing and able to provide written informed consent for the trial.
* Be male at birth and least 18 years of age on day of signing informed consent.
* Have measurable prostate cancer disease and be eligible for androgen deprivation therapy.
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function (all screening labs should be performed within 10 days of treatment initiation).
* Subjects have archival tumor tissue available or are willing to undergo a baseline biopsy prior to treatment.
* Subjects must have a life expectancy of at least 6 months.

Exclusion Criteria:

* Has an ECOG performance of 2 or higher.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the beginning of the treatment.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has a known allergy, intolerance, or medical contraindication to receiving the contrast dye required for the protocol-specified CT/MRI imaging
* Has any other medical intervention or condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives.
* Is not willing and able to provide written informed consent for the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | 3 years
  Feasibility of intermittent fasting (with the option of a plant-enriched diet) in prostate cancer patients receiving androgen deprivation therapy
Drop-out rate | 3 years
  Feasibility of intermittent fasting (with the option of a plant-enriched diet) in prostate cancer patients receiving androgen deprivation therapy

SECONDARY OUTCOMES:
Number of patients who achieve either partial or complete response by RECIST criteria on tumor imaging. | 3 years
  Clinical efficacy of the combination of intermittent fasting with or without a plant-enriched diet plus androgen deprivation therapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 3 years
  Safety, tolerability and reduction of common toxicities of the combination of intermittent fasting and the option of a plant-enriched diet intervention as compared to historical data.

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo/Great Lakes Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No